CLINICAL TRIAL: NCT03948594
Title: The Effect of Carbohydrate Loading on Gastric Residual Volume and Hunger Score: A Single Blind, Randomised Controlled Trial Study
Brief Title: The Effect of Carbohydrate Loading on Gastric Residual Volume and Hunger Score
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Bee Chen Lua, principal investigator, Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: USM/JEPeM/19010082
Record Dates: First submitted 2019-04-30; First posted 2019-05-14 (Actual); Last update posted 2019-05-17 (Actual); Status verified 2019-05

CONDITIONS: Gastric Residual Volume
Keywords: resource; gastric residual volume; hunger score
MeSH Terms: interventions — Health Resources

STUDY DESIGN:
Intervention Model Description: Subjects are randomised into 2 group: group A with 250cc plain water and group B with 1 packet resource(237ml)
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Allocation sequence is according computer generated random number list, it was prepared by an investigator with no clinical involvement in the trial. Allocation sequence was concealed from researcher enrolling and assessing participants. Allocation sequence will be sealed in sequentially numbered and opaque envelopes. A manila card will be placed inside envelop to render it impermeable to intense light. To prevent subversion of the allocation sequence, the name and I/C of the participant will be written on a book together with the series number on envelopes. The details in the book will be kept confidentially. After enrolled subject complete all baseline assessment, corresponding envelope will be enclosed by staff (who not involve in study) who prepare the drink. The staff need to ensure that the envelop still sealed when receive it. The staff will prepare the drink into identical container according to the assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- plain water (Placebo Comparator): subject drink 250cc plain water
  Interventions: Other: plain water
- resource (Active Comparator): subject drink 1 packet resource(237ml)
  Interventions: Dietary Supplement: resource

INTERVENTIONS:
Dietary Supplement: resource — 1 packet resource(237ml), 1.05kcal/ml, 53.6g carbohydrate and 9g protein
  Arms: resource
Other: plain water — 250ml plain water
  Arms: plain water

SUMMARY:
This study conducted is to assess effect of carbohydrate loading (maltodextrin with whey protein) to gastric volume 2 hours after ingestion via aspiration while doing OGDS (direct visualisation) and patient's wellbeing (hunger, thirst, weakness, tiredness, anxiety) for all patient planned for OGDS.

hypothesis H1: There is significant association between carbohydrate loading with residual gastric volume and subject's wellbeing H0: there is no significant association between carbohydrate loading with gastric residual volume and subject's wellbeing

DETAILED DESCRIPTION:
Patient scheduled for elective OGDS in HUSM from April 2019 to December 2019 with the complaint of one or more of the following symptoms: Bothersome postprandial fullness, early satiation, Epigastric pain or Epigastric burning are eligible to participate in the study. Patients who fulfilled exclusion criteria (History of upper gastrointestinal surgery, intestinal obstruction, patient with vomiting or mentally disable or who cannot give an informed consent) are ineligible.

If a patient fulfils the inclusion criteria, a suitable medical officer will discuss the trial with patient while reviewing patient in surgical outpatient clinic prior to OGDS. Patient will be approached again on the day of OGDS, if patient agree to participate in study, a written consent will be obtained. If patient refuse to participate in study, appropriate treatment and care still will be provided to patient. The consent form will provide information about the purpose of the study, the procedures to be followed, risks and benefits of participation. If patient agree to participate in the trial, subject will be enrolled in the study. Method of recruitment in this study is direct recruitment of potential study participants.

Stratified permuted block randomization was used. Randomization sequence was created using https://www.sealedenvelope.com/simple-randomiser/v1/lists and is stratified by gender (female and male) with 1:1 allocation. Random block sizes of 6 is used.

Allocation sequence is according computer generated random number list, it was prepared by an investigator with no clinical involvement in the trial. Allocation sequence was concealed from researcher enrolling and assessing participants. Allocation sequence will be sealed in sequentially numbered and opaque envelopes. A manila card will be placed inside envelop to render it impermeable to intense light. To prevent subversion of the allocation sequence, the name and I/C of the participant will be written on a book together with the series number on envelopes. The details in the book will be kept confidentially. After enrolled subject complete all baseline assessment, corresponding envelope will be enclosed by staff (who not involve in study) who prepare the drink. The staff need to ensure that the envelop still sealed when receive it. The staff will prepare the drink into identical container according to the assignment

Subjects are randomised into 2 group: group A with 250cc plain water and group B give 1 packet resource(237ml). Subjects need to finish the drink over 10minutes. After that, subjects are not allow to leave endoscope room before OGDS done to prevent consumption of other drink or food.

2 hours after that, subject undergo OGDS. OGDS is done follow standard protocol.

1. Patient lies in left lateral position
2. Medication to numb the back of throats (spray) will be given to prevent gagging during the passage of the instrument
3. A plastic mouth guard is placed between the teeth to prevent damage to the teeth and endoscope.
4. The endoscope (also called a gastroscope) will be inserted through the mouthpiece
5. A small container or yankauer suction is placed close to the mouth of a patient to collect saliva during and after the esophagogastroduodenoscopy
6. Endoscope will be inserted along the middle line of the soft palate.
7. Once endoscope advanced, patient may be asked to swallow to facilitate advancement of scope.
8. Throughout the procedure, no water flushing is allowed, only air inflation is allowed
9. visualised pooling of fluid in the stomach is aspirated until dry via direct visualization with endoscope. Aspirated fluid will be collected in suction reservoir and the fluid will be measured.

Subject's wellbeing is assessed via visual analogue scale (VAS) which consist of 5 parameters: hunger, thirst, anxiety, tiredness and weakness. Each scale consisted of ungraded, horizontal lines anchored at two ends. The left end of the scale represented "not at all" which score: 0 and the right end represented and "the most imaginable" which score: 100. Trained staff nurse will ask patient regarding level of 5 parameters and subject need to mark X somewhere along the horizontal line given before drink and before OGDS procedure.

All subjects are advised to inform assessor if there is adverse reaction. Medical personnel are available to manage any adverse events that might occur throughout the procedure.

The possible risk that may arise in the study include injury to the gastrointestinal's wall, aspiration and bleeding which is the similar risk for all patient going through OGDS procedure. Small volume of the drink will not cause psychological distress to subject, but its taste may not be palatable.

Sample size is calculated for all the objectives. However, the one that yield the biggest number is taken as the sample size.

objective 1 is to identify the gastric residual volume between subject with plain water (group A) and carbohydrate loading (group B). Sample size was calculated using comparing two means formula.

Objective 2 is to determined patient's well being for group A and group B. sample size was calculate using comparing paired difference formula.

For all sample size calculation, type I error was set at 5% (two tailed), Type 2 error was 20% (to achieve 80% power of study).

Corrected sample size is calculated after included 10% of dropout rate. Corrected sample size = calculated sample size/ (1-anticipated drop out rate).

After considering both objective, 1st objective give biggest number of sample size. Hence, 35 subject per group with a total number of 70 subjects are needed to study both objectives. after consider dropout rate, minimum sample size in this study is 39 subjects per group with a total number of 78 subjects.

The collected data will be entry and analyzed using SPSS version 24 (SPSS Inc., Chicago, IL, USA)

Objective 1 is to determine and compare gastric residual volume between group A and group B subjects. Independent T test is used to interpret the date.

Objective 2 is to determine and compare subject's well being before and after drink in between group A and group B. paired t test is used to determine effect of drink on subject's wellbeing before and after in each group. ANOVA is used to compare effect of the drink in both groups.

ELIGIBILITY:
Inclusion Criteria:

- Patient more than 18 years old

Exclusion Criteria:

* History of upper gastrointestinal surgery
* Intestinal obstruction
* Patient with vomiting
* Mentally disable or who cannot give an informed consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2019-05 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
gastric residual volume | 2 hours after plain water or carbohydrate loading
  Amount of gastric residual volume (ml) that has been aspirated via OGDS 2 hours after plain water or carbohydrate loading group

SECONDARY OUTCOMES:
patient's wellbeing | baseline (before drink) and 120minutes after drinking
  Subject's wellbeing is assessed via visual analogue scale (VAS) which consist of 5 parameters: hunger, thirst, anxiety, tiredness and weakness. Each scale consisted of ungraded, horizontal lines (with length of 100mm) anchored at two ends. The left end of the scale represented "not at all" which score: 0 and the right end represented and "the most imaginable" which score: 100. Subject need to mark X somewhere along the horizontal line given before drink and before OGDS procedure. Score of each parameter will be reported as mm.

CONTACTS AND LOCATIONS:
Overall Officials: Bee Chen Lua, M.D., Principal Investigator — USM surgery

REFERENCES:
- [Result] Adamina M, Kehlet H, Tomlinson GA, Senagore AJ, Delaney CP. Enhanced recovery pathways optimize health outcomes and resource utilization: a meta-analysis of randomized controlled trials in colorectal surgery. Surgery. 2011 Jun;149(6):830-40. doi: 10.1016/j.surg.2010.11.003. Epub 2011 Jan 14. PMID 21236454
- [Result] Asai T. Editorial II: Who is at increased risk of pulmonary aspiration? Br J Anaesth. 2004 Oct;93(4):497-500. doi: 10.1093/bja/aeh234. No abstract available. PMID 15361474
- [Result] Carmichael JC, Keller DS, Baldini G, Bordeianou L, Weiss E, Lee L, Boutros M, McClane J, Steele SR, Feldman LS. Clinical practice guideline for enhanced recovery after colon and rectal surgery from the American Society of Colon and Rectal Surgeons (ASCRS) and Society of American Gastrointestinal and Endoscopic Surgeons (SAGES). Surg Endosc. 2017 Sep;31(9):3412-3436. doi: 10.1007/s00464-017-5722-7. Epub 2017 Aug 3. No abstract available. PMID 28776285
- [Result] Dalal KS, Rajwade D, Suchak R. "Nil per oral after midnight": Is it necessary for clear fluids? Indian J Anaesth. 2010 Sep;54(5):445-7. doi: 10.4103/0019-5049.71044. PMID 21189883
- [Result] Faria MS, de Aguilar-Nascimento JE, Pimenta OS, Alvarenga LC Jr, Dock-Nascimento DB, Slhessarenko N. Preoperative fasting of 2 hours minimizes insulin resistance and organic response to trauma after video-cholecystectomy: a randomized, controlled, clinical trial. World J Surg. 2009 Jun;33(6):1158-64. doi: 10.1007/s00268-009-0010-x. PMID 19363695
- [Result] Gustafsson UO, Nygren J, Thorell A, Soop M, Hellstrom PM, Ljungqvist O, Hagstrom-Toft E. Pre-operative carbohydrate loading may be used in type 2 diabetes patients. Acta Anaesthesiol Scand. 2008 Aug;52(7):946-51. doi: 10.1111/j.1399-6576.2008.01599.x. Epub 2008 Mar 7. PMID 18331374
- [Result] Hausel J, Nygren J, Lagerkranser M, Hellstrom PM, Hammarqvist F, Almstrom C, Lindh A, Thorell A, Ljungqvist O. A carbohydrate-rich drink reduces preoperative discomfort in elective surgery patients. Anesth Analg. 2001 Nov;93(5):1344-50. doi: 10.1097/00000539-200111000-00063. PMID 11682427
- [Result] Helminen H, Viitanen H, Sajanti J. Effect of preoperative intravenous carbohydrate loading on preoperative discomfort in elective surgery patients. Eur J Anaesthesiol. 2009 Feb;26(2):123-7. doi: 10.1097/EJA.0b013e328319be16. PMID 19142085
- [Result] Hofman DL, van Buul VJ, Brouns FJ. Nutrition, Health, and Regulatory Aspects of Digestible Maltodextrins. Crit Rev Food Sci Nutr. 2016 Sep 9;56(12):2091-100. doi: 10.1080/10408398.2014.940415. PMID 25674937
- [Result] Kaska M, Grosmanova T, Havel E, Hyspler R, Petrova Z, Brtko M, Bares P, Bares D, Schusterova B, Pyszkova L, Tosnerova V, Sluka M. The impact and safety of preoperative oral or intravenous carbohydrate administration versus fasting in colorectal surgery--a randomized controlled trial. Wien Klin Wochenschr. 2010 Jan;122(1-2):23-30. doi: 10.1007/s00508-009-1291-7. PMID 20177856
- [Result] Kratzing C. Pre-operative nutrition and carbohydrate loading. Proc Nutr Soc. 2011 Aug;70(3):311-5. doi: 10.1017/S0029665111000450. PMID 21781358
- [Result] Nason KS. Acute Intraoperative Pulmonary Aspiration. Thorac Surg Clin. 2015 Aug;25(3):301-7. doi: 10.1016/j.thorsurg.2015.04.011. PMID 26210926
- [Result] Noblett SE, Watson DS, Huong H, Davison B, Hainsworth PJ, Horgan AF. Pre-operative oral carbohydrate loading in colorectal surgery: a randomized controlled trial. Colorectal Dis. 2006 Sep;8(7):563-9. doi: 10.1111/j.1463-1318.2006.00965.x. PMID 16919107
- [Result] Nygren J, Thorell A, Jacobsson H, Larsson S, Schnell PO, Hylen L, Ljungqvist O. Preoperative gastric emptying. Effects of anxiety and oral carbohydrate administration. Ann Surg. 1995 Dec;222(6):728-34. doi: 10.1097/00000658-199512000-00006. PMID 8526579
- [Result] Tran S, Wolever TM, Errett LE, Ahn H, Mazer CD, Keith M. Preoperative carbohydrate loading in patients undergoing coronary artery bypass or spinal surgery. Anesth Analg. 2013 Aug;117(2):305-13. doi: 10.1213/ANE.0b013e318295e8d1. Epub 2013 Jun 11. PMID 23757474
- [Derived] Lua BC, Md Hashim MN, Wong MS, Lee YY, Zakaria AD, Zakaria Z, Wan Zain WZ, Syed Abd Aziz SH, Yahya MM, Wong MP. Efficacy and safety of pre-gastroscopy commercial carbohydrate-rich whey protein beverage vs. plain water: a randomised controlled trial. Sci Rep. 2022 Oct 17;12(1):17355. doi: 10.1038/s41598-022-22363-1. PMID 36253448
- See also: Aspiration under anaesthesia: risk assessment and decision-making — http://dx.doi.org/10.1093/bjaceaccp/mkt053

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2019-04-15): https://cdn.clinicaltrials.gov/large-docs/94/NCT03948594/Prot_ICF_000.pdf